CLINICAL TRIAL: NCT04728854
Title: Improving Clinical Trial Recruitment and Outcome Measures in Bullous Pemphigoid
Brief Title: Telederm and Bullous Pemphigoid
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Ron Feldman, Assistant Professor, Emory University
Other Study IDs: STUDY00001274; 1R01AR076089-01A1 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult bullous pemphigoid patients: Patients with diagnosis of bullous pemphigoid will participate in monitoring with face to face assessment and remote telehealth visits with store and forward images captured.

SUMMARY:
The purpose of the study is to improve the quality of future clinical trials in bullous pemphigoid (BP), the investigators will monitor repeated measurement data from patients with BP on standard-of-care treatments at four week intervals for four months.

DETAILED DESCRIPTION:
The study team plans to recruit 45 subjects from the autoimmune blistering disease clinic at Emory Dermatology Clinic. The plan is to improve the quality of future clinical trials in bullous pemphigoid (BP), the team will monitor repeated measurement data from patients with BP on standard-of-care treatments at four week intervals for four months. This time frame will allow completion of both aims in the three year time period. Aim 1 will evaluate the BPDAI scoring over time with specific reductions in the activity score as future outcomes for therapeutic response and assess changes in patient reported outcomes particularly related to pruritus for future clinical trial endpoints. Aim 2 will focus on the development of teledermatology platform for improving patient recruitment and retention. The data from this proposal will be critical for future BP clinical trials and clarify gaps in the current knowledge related to the natural disease history of BP patients on standard-of-care therapies, changes in BPDAI scores over time, and pruritus specific outcome measures to define the quality of life impact.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > age 18
* Clinical and histological confirmation of bullous pemphigoid including at least subepidermal separation on H&E or a positive direct immunofluorescence along with indirect immunofluorescence which demonstrates staining to the roof on salt split skin or ELISA positivity for BP180 and/or BP230 autoantibodies
* Baseline BPDAI-TAS >5

Exclusion Criteria:

* Subjects who are unable to consent, language barriers, or other unspecified reason that in the opinion of the investigator makes the subject unsuitable for enrollment. Subjects that do not meet all of the enrollment criteria may not be enrolled. Any violations of these criteria must be reported in accordance with IRB Policies and Procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients from Emory Dermatology Clinic will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Change in Bullous pemphigoid disease area index (BPDAI) | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  Change in Bullous pemphigoid disease area index (BPDAI) activity score is the arithmetic sum of 3 subcomponents: cutaneous blisters/erosions, cutaneous urticaria/erythema, and mucosal blisters/erosions. Scores can range from 0 to 360 for BPDAI total activity (maximum 240 for total skin activity and 120 for mucosal activity), with higher scores indicating greater disease activity (worse outcome).

SECONDARY OUTCOMES:
Change in ItchyQol score | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  ItchyQoL focuses on pruritus as the main symptom impacting quality of life. ItchyQol score is based on an averaged 10-point visual analogue scale (VAS) over three time periods. Lower score correlates with better outcome.
Change in Autoimmune Bullous Disease Quality of Life score (ABQoL) | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  The Autoimmune Bullous Disease Quality of Life (ABQoL) score is a 17 item questionnaire assessing quality of life in patients with autoimmune blistering diseases. It is a patient reported score. Each question ranges from 0 to 3 points, with higher scores indicating poorer quality of life. The maximum ABQOL score is 51.
Change in Treatment of Autoimmune Bullous Disease Quality of Life (TABQoL) score | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  The Treatment of Autoimmune Bullous Disease Quality of Life (TABQoL) score is a patient reported score. The score is a 17 item questionnaire assessing quality of life in patients with autoimmune blistering diseases. Each question ranges from 0 to 3 points, with higher scores indicating poorer quality of life. The maximum TABQOL score is 51.
Change in patient and physician global assessment | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  The Physician and Patient Global Assessments will assess skin related health on a 0-5 scale at each visit. The lower score correlates with disease improvement (better outcome).
Number of participants with confidence that the dermatologist can help by looking at photos | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  This outcome is part of the patient satisfaction survey regarding teledermatology (TD) visits in order to encourage patient enrollment and retention for the length of the trial. Higher number of patients correlates with better outcome.
Number of participants with confidence that the teledermatology visit is more convenient than going to the dermatology clinic | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  This outcome is part of the patient satisfaction survey regarding teledermatology (TD) visits in order to encourage patient enrollment and retention for the length of the trial. Higher number of patients correlates with better outcome.
Number of participants that believe they will use the teledermatology service again | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  This outcome is part of the patient satisfaction survey regarding teledermatology (TD) visits in order to encourage patient enrollment and retention for the length of the trial. Higher number of patients correlates with better outcome.
Change in teledermatology satisfaction score | Baseline, monthly post-baseline for 4 months, 6 months post-baseline
  Teledermatology satisfaction will be evaluated using a survey that includes 3 questions. Possible score ranges from 0 to 3, with higher score correlating with better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Feldman, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Dermatology Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04728854/ICF_000.pdf